CLINICAL TRIAL: NCT07196267
Title: Combination Effect of Extracorporeal Shockwave and Cryoflow Therapy on Rotator Cuff Tendonitis in Stroke Patients
Brief Title: Shockwave and Cryoflow for Shoulder Pain After Stroke
Acronym: SW-CF-STROKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, reda abd elrazik, Associate Professor, Department of Physical Therapy for musculoskeletal disorders and its surgery, Faculty of Physical Therapy, Benha University, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT. BU. EC. Y
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Post-stroke Shoulder Pain,Rotator Cuff Tendonitis,Shoulder Spasticity
Keywords: Extracorporeal Shockwave Therapy; Cryoflow Therapy; Stroke Rehabilitation; Modified Ashworth Scale; Electromyography; Purdue Pegboard; Physical Therapy
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Weight-Bearing

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the Control Group (traditional PT + placebo) or the Experimental Group (traditional PT + real ESWT and Cryoflow). Both groups receive treatment concurrently over 8 weeks, with outcomes compared at baseline and post-intervention.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Traditional PT + Placebo (Placebo Comparator): Participants receive a traditional physical therapy program including stretching, strengthening, PNF, weight-bearing, and hand function training (Purdue Pegboard) for 40 minutes per session, 3 times per week for 8 weeks. Placebo extracorporeal shockwave and cryoflow therapy (device turned off or mimicked without active energy delivery) are applied to maintain blinding where possible.
  Interventions: Behavioral: Traditional Physical Therapy Program; Device: Placebo ESWT and Cryoflow
- Experimental: Traditional PT + ESWT + Cryoflow (Experimental): Participants receive the same traditional physical therapy program as the control group, plus active Extracorporeal Shockwave Therapy (7 Hz, 2.5-3 bar, 15 min) and Cryoflow Therapy (14°C, 15 min) applied sequentially before PT. Treatments are administered 3 times per week for 8 weeks.
  Interventions: Device: Extracorporeal Shockwave Therapy; Device: Cryoflow Therapy; Behavioral: Traditional Physical Therapy Program

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy — Delivered using Shock Master (Master Plus MP200, STORZ Medical AG, Switzerland). Applied at 7 Hz frequency, 2.5-3 bar pressure, for 15 minutes per session, 3 times per week for 8 weeks. Target: supraspinatus tendon region. Applied after Cryoflow therapy in experimental group.
  Other Names: ESWT
  Arms: Experimental: Traditional PT + ESWT + Cryoflow
Device: Cryoflow Therapy — Delivered using Cryoflow 1000IR (Model ICE-CT, EC). Applied at 14°C for 15 minutes per session, 3 times per week for 8 weeks. Applied directly over rotator cuff tendon region before ESWT in experimental group.
  Other Names: Cryoflow 1000IR
  Arms: Experimental: Traditional PT + ESWT + Cryoflow
Behavioral: Traditional Physical Therapy Program — tretching of shoulder flexors/adductors/internal rotators Strengthening of shoulder extensors/external rotators Weight-bearing exercises (sitting & quadruped) Neuromuscular Facilitation (PNF) for upper limb Hand dexterity training using Purdue Pegboard
  Other Names: Stretching, Strengthening, PNF, Weight-bearing, Hand Function Training
Device: Placebo ESWT and Cryoflow — Identical device setup as active ESWT and Cryoflow, but with energy delivery disabled (no acoustic pulses, no cold air output). Applied for 15 min each, mimicking active treatment to maintain blinding where possible. Used in control group alongside traditional PT.
  Other Names: Sham Shockwave ,Sham Cryoflow
  Arms: Control: Traditional PT + Placebo

SUMMARY:
This study aims to find out whether combining two physical therapy treatments - Extracorporeal Shockwave Therapy and Cryoflow Therapy - can help reduce shoulder pain and improve function in patients who have developed rotator cuff tendonitis after a stroke. Participants will be divided into groups to receive either one therapy alone or both therapies together. Researchers will measure pain levels, shoulder movement, and daily function before and after treatment to see which approach works best. The goal is to find a more effective, non-drug way to manage shoulder pain in stroke survivors and help them regain better use of their arm.

DETAILED DESCRIPTION:
This study will test whether combining Extracorporeal Shockwave Therapy (ESWT) and Cryoflow Therapy with traditional physical therapy is more effective than traditional therapy alone for reducing shoulder pain and improving arm function in stroke patients with rotator cuff tendonitis. Thirty stroke patients (ages 50-70) with moderate-to-severe shoulder spasticity (MAS grade 3) will be randomly assigned to one of two groups:

Group 1 (Control): Receives traditional physical therapy (stretching, strengthening, PNF, hand function training) + placebo ESWT/Cryoflow.

Group 2 (Experimental): Receives the same traditional therapy + real ESWT (7Hz, 15 min) and Cryoflow (14°C, 15 min).

All patients will be treated 3 times per week for 8 weeks. Before and after treatment, researchers will measure: shoulder muscle tone (Modified Ashworth Scale), range of motion (digital goniometer), muscle strength (tensiometer), hand dexterity (Purdue Pegboard), and muscle activity (electromyography). The goal is to find a better, non-drug way to relieve shoulder pain and restore function after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke confirmed by neurologist via physical examination and MRI. Age between 50 and 70 years. Moderate to severe shoulder spasticity, graded as Stage 3 on the Modified Ashworth Scale (MAS) for shoulder adductors.

Medically stable (vital signs within normal limits). Conscious, cooperative, and able to follow instructions. No orthopedic conditions, surgeries, or injuries affecting the shoulder or upper limb.

No sensory impairments (visual, auditory, proprioceptive) that would interfere with assessment or treatment.

Able to provide informed consent.

Exclusion Criteria:

* History of shoulder surgery or fracture. Presence of shoulder subluxation or dislocation. Severe cognitive impairment or inability to communicate. Uncontrolled hypertension, cardiac disease, or other unstable medical conditions.

Skin lesions, open wounds, or infection over the shoulder region. Diagnosis of frozen shoulder (adhesive capsulitis), rheumatoid arthritis, or other inflammatory joint diseases.

Previous treatment with ESWT or cryotherapy for shoulder within the last 6 months.

Use of botulinum toxin injections in the upper limb within the last 3 months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-10-10 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder Muscle Tone (Spasticity) | Baseline and after 8 weeks of treatment (24 sessions)
  Measured using the Modified Ashworth Scale (MAS) for shoulder adductors. MAS is a 6-point ordinal scale (0 = no increase in muscle tone, 5 = affected part rigid) to assess resistance during passive movement. Lower scores indicate reduced spasticity.

SECONDARY OUTCOMES:
Change in Shoulder Range of Motion | Baseline and after 8 weeks of treatment (24 sessions)
  Measured using a digital goniometer for active shoulder abduction and adduction. Range of motion recorded in degrees.
Change in Supraspinatus Muscle Strength | Baseline and after 8 weeks of treatment (24 sessions)
  Measured using a tensiometer (Lafayette, U.S.A.) to quantify isometric strength of the supraspinatus muscle. Force recorded in kilograms or Newtons.
Change in Hand Dexterity and Fine Motor Function | Baseline and after 8 weeks of treatment (24 sessions)
  Measured using surface electromyography (Neuropac apparatus) to record amplitude of motor unit action potentials (MUAP) of the supraspinatus muscle during standardized contractions. Reflects neuromuscular activation.
Change in Supraspinatus Muscle Electromyographic Activity | Baseline and after 8 weeks of treatment (24 sessions)
  Measured using surface electromyography (Neuropac apparatus) to record amplitude of motor unit action potentials (MUAP) of the supraspinatus muscle during standardized contractions. Reflects neuromuscular activation.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Benha University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided